CLINICAL TRIAL: NCT06671184
Title: Nomogram for Predicting Difficult Transoral and Submental Thyroidectomy
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Zhan, Doctor, Shanghai 6th People's Hospital
Other Study IDs: 2024-KY-236(K)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Differentiated thyroid cancer; Transoral and submental thyroidectomy; Surgical difficulty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult transoral and submental thyroidectomy: (1) operative time more than 75% of the overall study cases (2) severe intraoperative vascular or recurrent laryngeal nerve injury
  Interventions: Other: Observations on clinicopathological factors influencing the difficulty of surgery
- Normal transoral and submental thyroidectomy: the remaining of the entire study cases excluding the difficult cases
  Interventions: Other: Observations on clinicopathological factors influencing the difficulty of surgery

INTERVENTIONS:
Other: Observations on clinicopathological factors influencing the difficulty of surgery — Age, body mass index, gender, thyroid function parameters, lesion size, lesion location, ultrasound data

SUMMARY:
No prior studies have stratified the difficulty of transoral and submental thyroidectomy (TOaST). The investigators aimed to investigate preoperative factors as indicators of difficult TOaSTs and to develop a predictive model accordingly.

DETAILED DESCRIPTION:
Thyroid cancer is the most common endocrine malignancy, with a female predominance. Thyroidectomy is the main treatment for thyroid cancer, and considering the good prognosis of thyroid cancer, endoscopic thyroid surgery, which avoids neck incision, is being widely used in the clinic in order to improve the life treatment of patients. Among them, endoscopic thyroidectomy with transoral approach has a shorter learning curve because of the short surgical path. However, due to the complex structure of the neck, small space, and rich blood supply of the thyroid gland, surrounded by parathyroid glands and important nerves, endoscopic thyroid is difficult and has a long learning curve. In addition, a series of complications such as haemorrhage, hypoparathyroidism and laryngeal reentrant nerve injury can seriously affect the quality of patient survival. Difficult thyroidectomy is usually characterized by a long operative time, high intraoperative bleeding and a high incidence of postoperative complications. According to the literature, in open thyroid surgery, the degree of difficulty is associated with factors such as goiter, inflammation, and hyperthyroidism. However, the degree of difficulty of thyroidectomy due to various factors varies and is difficult to predict. Surgical difficulty is closely related to the outcome and safety of thyroidectomy, which is an urgent concern for surgeons. And there is no study on the degree of difficulty of transoral and submental endoscopic thyroidectomy, therefore, there is an urgent need for an effective and objective method to determine the preoperative factors affecting the degree of surgical difficulty and to establish a model for validation, so that it can be subsequently replicated in other hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of differentiated thyroid cancer with a maximum diameter not exceeding 4 cm
* Absence of suspicious lateral lymph nodes or distant metastases
* Participants with high cosmetic expectations
* Participants who underwent total thyroidectomy and central lymph node dissection.

Exclusion Criteria:

* Participants with fusion or fixation of lymph nodes in the neck
* Participants with history of neck surgery or radiation
* Participants with vocal fold fixation by preoperative fibrolaryngoscope
* Participants with preoperative examination suggestive of extrathyroidal invasion
* Participants with a significantly restricted neck

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with FNA proven differentiated thyroid cancer, were willing to undergo total thyroidectomy and central lymph node dissection via transoral and submental approach. Patients were well informed about the transoral and submental approach and were aware of the potential benefits and risks. Patient consented for us to use perioperative data.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrent laryngeal nerve injury | through study completion, an average of 1 year
  impaired vocal cord mobility confirmed by postoperative laryngoscopy
Number of participants with hypoparathyroidism | through study completion, an average of 1 year
  a postoperative parathyroid hormone level of less than 10 pg/ml
Number of participants with mental nerve injury | through study completion, an average of 1 year
  a postoperative numbness in the lower lip and submental area
operative time | through study completion, an average of 1 year
  operative time was defined as the duration from incision to closure, and was collected from anesthesia record sheet

SECONDARY OUTCOMES:
hospitalization | through study completion, an average of 1 year
  days of hospitalization
degree of pain | approximately 4 hours after surgery and on postoperative day 1
  pain intensity was assessed using a standard visual analogue score, with a score of 0 to 10 corresponding to no pain to the most severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhan, Doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data are available on request due to privacy or other restrictions. The data that support the findings of this study are available on request from Ling Zhan. The data are not publicly available due to them containing information that could compromise research participant privacy.

REFERENCES:
- [Result] Zhan L, Xuan M, Ding H, Liang J, Zhao Q, Chen L, Yang Z, Cheng X, Kuang J, Yan J, Cai W, Qiu W. Learning curve of trans-areola single-site endoscopic thyroidectomy in a high-volume center: A CUSUM-based assessment. Cancer Med. 2023 Aug;12(16):16846-16858. doi: 10.1002/cam4.6307. Epub 2023 Jul 3. PMID 37395126
- [Result] Liang J, Zhan L, Xuan M, Zhao Q, Chen L, Yan J, Kuang J, Tan J, Qiu W. Thyroidectomy for thyroid cancer via transareola single-site endoscopic approach: results of a case-match study with large-scale population. Surg Endosc. 2022 Feb;36(2):1394-1406. doi: 10.1007/s00464-021-08424-y. Epub 2021 Mar 29. PMID 33782758